CLINICAL TRIAL: NCT05824728
Title: Clinical Trial Evaluating the Efficacy and Safety of AGB101 for Treatment of Parkinson's Disease Related Psychosis
Acronym: AGB101 PDP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: AgeneBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00318189
Record Dates: First submitted 2023-04-06; First posted 2023-04-24 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease Psychosis
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AGB101 first, then placebo (Experimental): AGB101 (low-dose levetiracetam, 220 mg, extended release tablet) once daily for 6 weeks, washout (4 weeks), then placebo capsule once daily for 6 weeks.
  Interventions: Drug: AGB101
- placebo first, then AGB101 (Experimental): Placebo capsule once daily for 6 weeks, washout (4 weeks), then AGB101 (low-dose levetiracetam, 220 mg, extended release tablet) once daily for 6 weeks.
  Interventions: Drug: AGB101

INTERVENTIONS:
Drug: AGB101 — low-dose levetiracetam, 220 mg, extended release tablet
  Other Names: levetiracetam

SUMMARY:
This clinical trial will test whether AGB101 (low-dose levetiracetam, 220 mg, extended release tablet) can improve symptoms of psychosis in Parkinson's disease. Participants will be asked to complete up to 5 in-person study visits over approximately 20 weeks. Participants will receive both AGB101 and a placebo to take once a day for 6 weeks, with a 4-week washout in between. Participation will also involve physical/neurological exams, questionnaires, paper and pencil tests, providing blood and urine samples, and completing two MRI exams.

DETAILED DESCRIPTION:
Hallucinations and memory impairment have a parallel clinical course in Parkinson's disease (PD) and are independently associated dysfunction and pathology accumulation in hippocampal subregions. Similar alterations of hippocampal function are found in schizophrenic patients with memory impairment and positive psychotic symptoms. These findings suggest that dysfunction of the hippocampus may be a shared mechanism for memory impairment and psychosis across diseases. This investigation aims to address these questions and assess the efficacy of AGB101 for the treatment of psychosis in PD.

ELIGIBILITY:
Subjects must meet all of the following inclusion criteria at screening:

1. Subjects between 40 and 85 years old (inclusive) in good general health:

   1. Willing and able to consent and participate for the duration of the study.
   2. Have eighth-grade education or good work history sufficient to exclude mental retardation.
   3. Have visual and auditory acuity adequate for neuropsychological testing.
   4. Have proficient fluency of the native local language to participate in all the neuropsychological test assessments.
2. Have a study partner who has sufficient contact (≥ 2 hours per week) with the subject to assist with dosing of study medication (if necessary) and provide assessments of any changes and an independent evaluation of the subject's functioning.
3. Have PDP as defined by all of the following criteria and consistent with the National Institute of Neurological Disorders and Stroke/National Institute of Mental Health (NINDS/NIMH) criteria:

   1. Meets United Kingdom brain bank criteria for PD
   2. Presence of at least one of the following symptoms

      * Illusions
      * False sense of presence
      * Hallucinations
      * Delusions
   3. The symptoms of Criterion b occur after the onset of PD.
   4. The symptoms of Criterion b are recurrent or continuous for 1 month.
   5. The symptoms of Criterion b are not better accounted for by another cause of Parkinsonism such as dementia with Lewy bodies, psychiatric disorders such as schizophrenia, schizoaffective disorder, delusional disorder, or mood disorder with psychotic features, or a general medical condition including delirium.
   6. May have the following associated features:

      * With/without insight
      * With/without dementia
      * With/without treatment for PD
4. Patients must be experiencing symptom(s) of Criterion 3b at least once a week during the 4 weeks prior to the screening visit.
5. Patients being treated for symptom(s) of Criterion 3b must be off medication for at least 2 weeks prior to randomization.
6. Patients must be on a stable regimen of medication for PD for at least 4 weeks prior to randomization.
7. Permitted medications:

   1. With potential pro-cognitive effects, such as cholinesterase inhibitors, memantine, estrogen replacement therapy, must be at a stable dose for 1 month prior to screening and expected to remain stable throughout the study
   2. Antidepressants must be at a stable dose for 1 month prior to screening and expected to remain stable throughout the study.
   3. Antipsychotics must be must be at a stable dose for 1 month prior to screening and expected to remain stable throughout the study.
8. Willing and able to undergo repeated MRI scans (3 Tesla) with no contraindications to MRI.
9. Participant and partner must both be willing to use an effective contraception for duration of the study and for 4 days after it. For women, effective contraception may be hormonal; for men, a condom.

Exclusion Criteria:

Subjects must not meet any of the following exclusion criteria at screening:

1. Use of anticonvulsant medications within 1 month prior to the baseline visit.
2. Participation in a therapeutic clinical study for any medical or psychiatric indications within 1 month of the screening visit, or at any time during the study. Subjects must understand that they may only enroll in this clinical study once; they may not enroll in any other clinical study while participating in the current study, and they may not participate in a clinical study of a drug, biologic, therapeutic device, or medical food, in which the last dose/administration was received within 1 month prior to screening.
3. History of hypersensitivity or lack of tolerability to AGB101 (levetiracetam).
4. Severe renal impairment (creatinine clearance of < 30 mL/minute) or undergoing hemodialysis.
5. Delirium due to the presence of an acute metabolic encephalopathy secondary to infection or from any other cause as assessed by the investigator based on labs, history, and physical exam.
6. Neurological disorder other than Parkinson's disease, such as Alzheimer's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder (lifetime history; infant febrile seizures are not exclusionary), subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits, or known structural brain abnormalities, that in the opinion of the investigator might interfere with the conduct of the study.
7. Prior diagnosis of schizophrenia, bipolar disorder or other psychotic disorder other than PD-related psychosis.
8. Stereotactic surgery for deep brain stimulation (DBS), presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body that constitute a contraindication to having an MRI scan.
9. History of alcohol or substance abuse or dependence within the past 3 years (DSM-5 criteria).
10. Any significant systemic illness or unstable medical condition that could lead to difficulty in complying with the protocol requirements.
11. Any unstable medical condition that is likely to require new medical or surgical treatment during the course of the study and where such treatments might affect the collection of efficacy data.
12. Unable or unwilling to provide informed consent or to comply with study procedures.
13. Patient or caregiver unable to administer daily oral dosing of study drug.
14. Current suicidal ideation.
15. Female subjects must not be pregnant or lactating.
16. Any other reason, which in the opinion of the investigator would confound proper interpretation of the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in hallucinations/delusions as assessed by the Enhanced Scale for Assessment of Positive Symptoms in Parkinson's Disease (eSAPS-PD) | Screening, Baseline, Week 3, Week 6, Week 13, Week 16
  The eSAPS-PD is used to track changes in hallucinations and other psychotic symptoms over time. It was adapted from the scale for the assessment of positive symptoms (SAPS), which is used to track positive symptoms in patients with schizophrenia. The eSAPS-PD is a 13-item questionnaire which specifically assesses the frequency or severity of the most common types of hallucinations or delusions found in PD, namely auditory hallucinations, voices conversing, somatic or tactile hallucinations, visual hallucinations, persecutory delusions, delusions of jealousy and delusions of reference. In addition, the enhanced version assesses minor psychotic phenomena such as illusions, passage hallucinations, and presence hallucinations. Each item is rated from 0-5, with 0 representing none and 5 representing severe and frequent symptoms, and the total score ranges from 0 to 65.

SECONDARY OUTCOMES:
Change in hippocampal overactivity as measured by fMRI (functional Magnetic Resonance Imaging) | Week 6, Week 16
  The secondary efficacy evaluation is confirmation of target engagement demonstrated by reduction in hippocampal overactivity comparing the end of the active treatment period compared to the end of the placebo treatment condition as measured by task-based functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Bakker, Ph.D., Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No